CLINICAL TRIAL: NCT03336541
Title: Effects of Intraoperative Low-dose Ketamine on Incidence of Postpartum Depression in Parturients With Prenatal Depression Undergoing Cesarean Delivery: Blind Test, Randomized, Placebo-controlled Trial
Brief Title: Low-dose Ketamine and Postpartum Depression in Parturients With Prenatal Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017[36]
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Perinatal Depression; Ketamine; Cesarean Delivery; Postpartum Depression
Keywords: Prenatal depression; Ketamine; Cesarean delivery; Postpartum depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine group (Experimental): Low-dose ketamine (0.5 mg/kg in 100 ml normal saline) is intravenously infused in 40 minutes after childbirth during cesarean delivery.
  Interventions: Drug: Ketamine
- Placebo group (Placebo Comparator): Placebo (100 ml normal saline) is intravenously infused in 40 minutes after childbirth during cesarean delivery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine (0.5 mg/kg in 100 ml normal saline) will be administered by intravenous infusion in 40 minutes after childbirth during cesarean delivery.
  Other Names: Ketamine hydrochloride
  Arms: Ketamine group
Drug: Placebo — Placebo (100 ml normal saline) will be administered by intravenous infusion in 40 minutes after childbirth during cesarean delivery.
  Other Names: Normal saline
  Arms: Placebo group

SUMMARY:
Postpartum depression is common in mothers early after childbirth and produces harmful effects not only on mothers, but also on infants and young children. Parturients with prenatal depression are at increased of postpartum depression. Low-dose ketamine can be used for antidepressant therapy. We hypothesize that low-dose ketamine has a therapeutic effect on parturients with prenatal depression. This study is designed to investigate whether low-dose ketamine administered during cesarean delivery can decrease the incidence of postpartum depression in parturients with prenatal depression.

DETAILED DESCRIPTION:
Postpartum depression refers to maternal depression developed early after childbirth, with reported incidences varied from 15% to 20%. The development of postpartum depression produces harmful effects not only on mothers, but also on infants and young children. Prenatal depression or high depression score is an independent risk factor for the development of postpartum depression.

Ketamine is commonly used as an general anesthetic. In addition, low-dose ketamine is recommended for antidepressant therapy. We hypothesize that low-dose ketamine has a therapeutic effect on parturients with prenatal depression. However, evidences in this aspect are insufficient. The purpose of this study is to investigate whether low-dose ketamine administered during cesarean delivery can decrease the incidence of postpartum depression in parturients with prenatal depression.

ELIGIBILITY:
Inclusion Criteria:

* Parturients with age from 18 to 45 years and scheduled for elective cesarean delivery;
* Prenatal depression score (EPDS) of 10 or higher;
* Provide written informed consents.

Exclusion Criteria:

* Refused to participate in the study;
* History of schizophrenia or other disease that prevent normal communication before delivery;
* Presence of contraindications to neuraxial anesthesia, including central nervous system diseases (such as poliomyelitis), spinal diseases (such as spinal canal tumor, lumbar disc prolapse, history of spinal trauma), systemic infection (such as sepsis, bacteremia), local infection in the site of puncture, or coagulopathy;
* Severe complications during pregnancy (such as severe preeclampsia, placenta accreta, HELLP syndrome);
* Severe comorbidity before pregnancy (such as severe cardiac dysfunction);
* Scheduled to undergo cesarean delivery under general anesthesia;
* Other reasons that are considered unsuitable for study participation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
The score of postpartum depression at 48 hous after childbirth. | At 48 hours after delivery.
  Postpartum depression is assessed with Edinburgh postnatal depression scale (EPDS) at 48 hours after childbirth. The EPDS is a 10-item self-rating post-natal depression scale. Each item is scored from 0 to 3, resulting an overall score ranging from 0-30; a high score indicates severe depression.

SECONDARY OUTCOMES:
Time of first breast feeding. | From delivery to 24 hours after delivery.
  Time of first breast feeding.
The proportion of neonates with breast feeding. | At 24 hours after delivery.
  The proportion of neonates with breast feeding.
Duration of neonatal sleep within 24 hours after delivery. | During the first 24 hours after delivery.
  Duration of neonatal sleep within 24 hours after delivery.
Length of stay in hospital after delivery. | From childbirth up to 30 days after delivery.
  Length of stay in hospital after delivery.
The score of postpartum depression at 42 days after delivery. | At 42 days after delivery.
  Postpartum depression is assessed with EPDS at 42 days after childbirth.
Incidence of postpartum depression at 42 days after delivery. | At 42 days after delivery.
  Postpartum depression is assessed with EPDS at 42 days after childbirth. A EPDS score of 10 or above is defined as postpartum depression.
Incidence of maternal complications with 42 days after delivery. | From childbirth up to 42 days after delivery.
  Incidence of maternal complications with 42 days after delivery.
Incidence of neonatal complications with 42 days after delivery. | From childbirth up to 42 days after delivery.
  Incidence of neonatal complications with 42 days after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel M, Bailey RK, Jabeen S, Ali S, Barker NC, Osiezagha K. Postpartum depression: a review. J Health Care Poor Underserved. 2012 May;23(2):534-42. doi: 10.1353/hpu.2012.0037. PMID 22643605
- [Background] Stein A, Pearson RM, Goodman SH, Rapa E, Rahman A, McCallum M, Howard LM, Pariante CM. Effects of perinatal mental disorders on the fetus and child. Lancet. 2014 Nov 15;384(9956):1800-19. doi: 10.1016/S0140-6736(14)61277-0. Epub 2014 Nov 14. PMID 25455250
- [Background] Verbeek T, Bockting CL, van Pampus MG, Ormel J, Meijer JL, Hartman CA, Burger H. Postpartum depression predicts offspring mental health problems in adolescence independently of parental lifetime psychopathology. J Affect Disord. 2012 Feb;136(3):948-54. doi: 10.1016/j.jad.2011.08.035. Epub 2011 Sep 17. PMID 21930302
- [Background] Feldman R, Granat A, Pariente C, Kanety H, Kuint J, Gilboa-Schechtman E. Maternal depression and anxiety across the postpartum year and infant social engagement, fear regulation, and stress reactivity. J Am Acad Child Adolesc Psychiatry. 2009 Sep;48(9):919-927. doi: 10.1097/CHI.0b013e3181b21651. PMID 19625979
- [Background] Kersten-Alvarez LE, Hosman CM, Riksen-Walraven JM, van Doesum KT, Smeekens S, Hoefnagels C. Early school outcomes for children of postpartum depressed mothers: comparison with a community sample. Child Psychiatry Hum Dev. 2012 Apr;43(2):201-18. doi: 10.1007/s10578-011-0257-y. PMID 22011810
- [Background] Raposa E, Hammen C, Brennan P, Najman J. The long-term effects of maternal depression: early childhood physical health as a pathway to offspring depression. J Adolesc Health. 2014 Jan;54(1):88-93. doi: 10.1016/j.jadohealth.2013.07.038. Epub 2013 Sep 20. PMID 24060574
- [Background] Naicker K, Wickham M, Colman I. Timing of first exposure to maternal depression and adolescent emotional disorder in a national Canadian cohort. PLoS One. 2012;7(3):e33422. doi: 10.1371/journal.pone.0033422. Epub 2012 Mar 26. PMID 22461893
- [Background] Schiller CE, Meltzer-Brody S, Rubinow DR. The role of reproductive hormones in postpartum depression. CNS Spectr. 2015 Feb;20(1):48-59. doi: 10.1017/S1092852914000480. Epub 2014 Sep 29. PMID 25263255
- [Background] Hart AR, Farber KG, Kellner ChH. Postpartum Depression. N Engl J Med. 2017 Mar 2;376(9):895. doi: 10.1056/NEJMc1616547. No abstract available. PMID 28252268
- [Background] Kingston D, McDonald S, Austin MP, Tough S. Association between Prenatal and Postnatal Psychological Distress and Toddler Cognitive Development: A Systematic Review. PLoS One. 2015 May 21;10(5):e0126929. doi: 10.1371/journal.pone.0126929. eCollection 2015. PMID 25996151
- [Background] Layer RT, Popik P, Olds T, Skolnick P. Antidepressant-like actions of the polyamine site NMDA antagonist, eliprodil (SL-82.0715). Pharmacol Biochem Behav. 1995 Nov;52(3):621-7. doi: 10.1016/0091-3057(95)00155-p. PMID 8545484
- [Background] Meloni D, Gambarana C, De Montis MG, Dal Pra P, Taddei I, Tagliamonte A. Dizocilpine antagonizes the effect of chronic imipramine on learned helplessness in rats. Pharmacol Biochem Behav. 1993 Oct;46(2):423-6. doi: 10.1016/0091-3057(93)90374-3. PMID 7903459
- [Background] Moryl E, Danysz W, Quack G. Potential antidepressive properties of amantadine, memantine and bifemelane. Pharmacol Toxicol. 1993 Jun;72(6):394-7. doi: 10.1111/j.1600-0773.1993.tb01351.x. PMID 8361950
- [Background] Papp M, Moryl E. Antidepressant activity of non-competitive and competitive NMDA receptor antagonists in a chronic mild stress model of depression. Eur J Pharmacol. 1994 Sep 22;263(1-2):1-7. doi: 10.1016/0014-2999(94)90516-9. PMID 7821340
- [Background] Przegalinski E, Tatarczynska E, Deren-Wesolek A, Chojnacka-Wojcik E. Antidepressant-like effects of a partial agonist at strychnine-insensitive glycine receptors and a competitive NMDA receptor antagonist. Neuropharmacology. 1997 Jan;36(1):31-7. doi: 10.1016/s0028-3908(96)00157-8. PMID 9144639
- [Background] Trullas R, Skolnick P. Functional antagonists at the NMDA receptor complex exhibit antidepressant actions. Eur J Pharmacol. 1990 Aug 21;185(1):1-10. doi: 10.1016/0014-2999(90)90204-j. PMID 2171955
- [Background] Sanacora G, Gueorguieva R, Epperson CN, Wu YT, Appel M, Rothman DL, Krystal JH, Mason GF. Subtype-specific alterations of gamma-aminobutyric acid and glutamate in patients with major depression. Arch Gen Psychiatry. 2004 Jul;61(7):705-13. doi: 10.1001/archpsyc.61.7.705. PMID 15237082
- [Background] Sanacora G, Zarate CA, Krystal JH, Manji HK. Targeting the glutamatergic system to develop novel, improved therapeutics for mood disorders. Nat Rev Drug Discov. 2008 May;7(5):426-37. doi: 10.1038/nrd2462. PMID 18425072
- [Background] McCullumsmith RE, Kristiansen LV, Beneyto M, Scarr E, Dean B, Meador-Woodruff JH. Decreased NR1, NR2A, and SAP102 transcript expression in the hippocampus in bipolar disorder. Brain Res. 2007 Jan 5;1127(1):108-18. doi: 10.1016/j.brainres.2006.09.011. Epub 2006 Nov 17. PMID 17113057
- [Background] Paul IA, Nowak G, Layer RT, Popik P, Skolnick P. Adaptation of the N-methyl-D-aspartate receptor complex following chronic antidepressant treatments. J Pharmacol Exp Ther. 1994 Apr;269(1):95-102. PMID 8169857
- [Background] Boyer PA, Skolnick P, Fossom LH. Chronic administration of imipramine and citalopram alters the expression of NMDA receptor subunit mRNAs in mouse brain. A quantitative in situ hybridization study. J Mol Neurosci. 1998 Jun;10(3):219-33. doi: 10.1007/BF02761776. PMID 9770644
- [Background] Aan Het Rot M, Zarate CA Jr, Charney DS, Mathew SJ. Ketamine for depression: where do we go from here? Biol Psychiatry. 2012 Oct 1;72(7):537-47. doi: 10.1016/j.biopsych.2012.05.003. Epub 2012 Jun 16. PMID 22705040
- [Background] DiazGranados N, Ibrahim LA, Brutsche NE, Ameli R, Henter ID, Luckenbaugh DA, Machado-Vieira R, Zarate CA Jr. Rapid resolution of suicidal ideation after a single infusion of an N-methyl-D-aspartate antagonist in patients with treatment-resistant major depressive disorder. J Clin Psychiatry. 2010 Dec;71(12):1605-11. doi: 10.4088/JCP.09m05327blu. Epub 2010 Jul 13. PMID 20673547
- [Background] Katalinic N, Lai R, Somogyi A, Mitchell PB, Glue P, Loo CK. Ketamine as a new treatment for depression: a review of its efficacy and adverse effects. Aust N Z J Psychiatry. 2013 Aug;47(8):710-27. doi: 10.1177/0004867413486842. Epub 2013 May 9. PMID 23661785
- [Derived] Wang S, Deng CM, Zeng Y, Ma JH, Qu Y, Wang DX. Single low-dose ketamine infusion for women with prenatal depressive symptoms undergoing cesarean delivery: A pilot randomized trial. Front Surg. 2022 Dec 8;9:1050232. doi: 10.3389/fsurg.2022.1050232. eCollection 2022. PMID 36570810